CLINICAL TRIAL: NCT06563453
Title: Implication of Cognitive Reserve in Non-pharmacological Intervention Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: NU21-04-00652
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2023-12

CONDITIONS: Aging; Mild Cognitive Impairment; Dementia With Lewy Bodies
MeSH Terms: conditions — Cognitive Dysfunction; Lewy Body Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- sham stimulation (Sham Comparator): Two inactive electrodes (anodes and cathodes) - placed over Medial frontal lobe and Inferior parietal lobe. The flow of current discontinues after 20 seconds, the stimulation continues.
  Interventions: Device: transcranial alternating current stimulation
- frontal stimulation (Experimental): One active electrode (anode and cathode) - placed over Medial frontal lobe, one inactive electrode (anode and cathode) - placed over Inferior parietal lobe.
  Current intensity - 2 (milliamperes) mA, frequency: theta 4.51 Hz, stimulation time: 20 minutes
  Interventions: Device: transcranial alternating current stimulation
- frontoparietal stimulation (Experimental): One active electrode (anode and cathode) - placed over Medial frontal lobe, another active electrode (anode and cathode) - placed over Inferior parietal lobe.
  Current intensity - 2 mA, frequency: theta 4.51 Hz in-phase, stimulation time: 20 minutes
  Interventions: Device: transcranial alternating current stimulation

INTERVENTIONS:
Device: transcranial alternating current stimulation — Transcranial Alternating Current Stimulation (tACS) is a tool that administers a weak alternating current (in the range of 0.1 to 4 mA), most often with a sinusoidal waveform, between electrodes placed over target areas. This can entrain the subjacent neuronal networks favouring the firing at specific frequencies of interest, in certain cases, with effects outlasting the stimulation duration up to 70 min.

SUMMARY:
Cognitive reserve (CR) is defined as the gradual accumulation of neural resources and their adaptability (i.e., efficiency, capacity, flexibility) due to genetic and/or lifelong environmental factors that mitigate the cognitive effects of age-related processes and brain diseases. Transcranial alternating current stimulation (tACS) can be used to entrain underlying neuronal networks, promoting firing at specific frequencies. Recent studies have demonstrated that fronto-parietal theta oscillatory activity entrainment via tACS leads to working memory enhancement in healthy subjects. However, there remains significant variability in stimulation-induced aftereffects across individuals.

Emerging literature suggests that individual differences, such as CR levels, may be crucial in predicting the benefits of treatment interventions, as they reflect available neural capacity and flexibility. A novel interventional approach is proposed to study CR, utilizing both conventional static proxies, such as premorbid intellect and educational attainment, and dynamic markers, including pupillometry, resting-state, and task-induced functional MRI. By employing cutting-edge noninvasive brain stimulation (NIBS) techniques, the study will acutely modulate network properties to examine the influence of CR on immediate cognitive and brain functional aftereffects induced by the intervention. In addition to focusing on cognitively healthy older adults, this study will, for the first time, include patients with mild cognitive impairment with Lewy bodies (MCI-LB), a prodromal stage of the second most common degenerative dementia after Alzheimer's disease.

DETAILED DESCRIPTION:
A novel interventional approach is proposed for studying cognitive reserve (CR) using dynamic biomarkers, including:

Neuromelanin-sensitive MRI sequences to evaluate signal intensity of the locus coeruleus, Resting-state functional MRI (rs-fMRI) to evaluate network properties such as modularity and local and global efficiency, Baseline dynamic rs-fMRI to evaluate mean dwell time and number of transitions between states, and Baseline task-induced activation to evaluate engagement of "domain-specific" and "domain-general" regions during the 'offline' transfer working memory (WM) task performance, i.e., tasks solved after transcranial alternating current stimulation (tACS).

These dynamic biomarkers are used in addition to established conventional static proxies (education and premorbid intellect).

Specifically, the study aims to:

Assess which CR biomarkers and conventional CR proxies, alone or in combination, best predict the tACS-induced magnitude of cognitive enhancement of the 'online' WM task (solved while stimulated).

Evaluate the influence of CR on the recruitment of compensatory mechanisms (as assessed by task-induced fMRI and rs-fMRI) induced by tACS for solving challenging WM tasks.

Investigate how the CR level moderates the relationship between the magnitude and spatial patterns of brain flexibility changes induced by an acute tACS (as measured by pupil dilation during the online WM task performance and pre-post tACS resting-state functional connectivity changes within and between large-scale brain networks) and cognitive tACS-induced enhancement (as measured by 'online' WM task performance and changes in the 'offline' transfer task performance solved after stimulation).

ELIGIBILITY:
Inclusion Criteria:

1. Intact cognitive performance as assessed by cognitive evaluation.
2. Subjects with possible or probable mild cognitive impairment with Lewy bodies (MCI-LB).

Exclusion Criteria:

Presence of dementia as assessed by a cognitive test battery and evaluation of daily activities.

Any major psychiatric disorder. History of neurological disease affecting the central nervous system (e.g., tumor, epilepsy, stroke, etc.).

Severe or repeated head injury. Non-compensated internal or oncological disease. MRI-incompatible metal in the body (e.g., pacemaker). Left-handedness.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy and reaction times of the visual N-back task in tACS conditions:tACS conditions | 3.5 years
  'Online' working memory (WM) task accuracy and reaction times (RT) in both active and sham tACS conditions.
  tACS conditions
Accuracy and reaction times of the verbal N-back task in tACS conditions: tACS conditions | 3.5 years
  'Offline' WM task accuracy and reaction times (RT) in both active and sham tACS conditions.
  tACS conditions

SECONDARY OUTCOMES:
Cognitive reserve moderator: | 3.5 years
  Identification of which cognitive reserve proxies or indexes are most effective at moderating tACS-induced changes.
tACS-induced functional connectivity changes: | 3.5 years
  tACS-induced neural changes, including resting-state functional connectivity (rs-FC) within and between large-scale brain networks, dynamic rs-fMRI measures, and task-induced BOLD (Blood-Oxygen-Level Dependent) signal increases assessed at baseline and immediately after each stimulation.
Pupillary changes | 3.5
  Measures of pupil dilation during the N-back task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Eliášová, Ph.D., Principal Investigator — Masaryk University
Locations (1):
- CEITEC Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No
available upon reasonable request

REFERENCES:
- [Derived] Mitterova K, Pupikova M, Gajdos M, Eliasova I, Rektorova I. Optimizing tACS for working memory: differential outcomes in healthy aging and non-amnestic mild cognitive impairment. Alzheimers Res Ther. 2025 Dec 2;18(1):2. doi: 10.1186/s13195-025-01922-4. PMID 41331881